CLINICAL TRIAL: NCT03336086
Title: Reduction of Natural Killer Cell (CD16/56) and T-lymphocyte (CD3) Subset Counts After a Weight Loss Program Using Anti-obesity Drugs in Obese Women: a Non-randomized Controlled Trial
Brief Title: Effect of Weight Reduction on Immunity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mahsa Mehrdad, Principal investigator, Shiraz University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 900413
Record Dates: First submitted 2017-09-17; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Lymphocytes; Weight Loss; Viral Diseases; Immunity; Anti-obesity Agents
MeSH Terms: conditions — Weight Loss; Virus Diseases | interventions — Weight Reduction Programs

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- experimental (Other): This group underwent a weight loss program
  Interventions: Combination Product: weight loss program
- control (No Intervention): This group underwent adlibitum diet + physical activity

INTERVENTIONS:
Combination Product: weight loss program — A low calorie diet+ Orlistat+ Soluble Fiber+ Physical activity
  Other Names: experimental
  Arms: experimental

SUMMARY:
This study included two groups of premenopausal healthy obese women. Experimental group underwent a weight loss program involved a low calorie diet plus anti-obesity drugs and moderate physical activity and control group underwent an ad libitum diet. At baseline and after a 10-15% weight loss lymphocyte subgroups were analyzed and compared between two group.

DETAILED DESCRIPTION:
TCD3 and NKC CD16/56 were decreased significantly. Hence this weight loss program impaired viral immunity

ELIGIBILITY:
Inclusion Criteria:

* BMI >=30
* female
* healthy
* no smoking
* not lactating
* not pregnant
* no medication use

Exclusion Criteria:

* pregnancy
* any disease
* any medication use
* iron and zinc deficiency
* any supplement use

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2012-03-20 (Actual); Primary Completion 2012-11-30 (Actual); Study Completion 2012-12-25 (Actual)

PRIMARY OUTCOMES:
lymphocyte subgroups | 6 months
  TCD3. TCD4. TCD8. BCD19. NKCs CD16/56 (Cells/microliter) by flowcytometry

SECONDARY OUTCOMES:
Body Mass Index | 6 months
  (Kg/m^2) by equation
Biomarkers | 6 months
  ZN, Iron (microgram/deciliter) by biochemical assessment
Systolic blood pressure | 6 months
  (mmHg) by manometer
diastolic blood pressure | 6 months
  (mmHg) by manometer
Weight | 6 months
  (Kg) by Bioelectric impedance analyser
Fat Mass | 6 months
  (Kg) by Bioelectric impedance analyser
Fat Free Mass | 6 months
  (Kg) by Bioelectric impedance analyser
Trunk Fat | 6 months
  (Kg) by Bioelectric impedance analyser
Waist circumference | 6 months
  (cm) by meter tape